CLINICAL TRIAL: NCT03698214
Title: Is There a Worse Outcome When the Systolic Blood Pressure is Lower Than Heart Rate in Those Adult Trauma Patients With Isolated Head/Neck Injury
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CGRPG8F0011
Record Dates: First submitted 2018-10-02; First posted 2018-10-05 (Actual); Last update posted 2018-10-05 (Actual); Status verified 2016-03

CONDITIONS: Traumatic Brain Injury
Keywords: systolic blood pressure; reversed shock index; traumatic brain injury; mortality
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- isolated traumatic brain injury: Adult patients having isolated traumatic brain injury with a head abbreviated injury scale (AIS) ≥ 3 and without severe injury to other regions (other AIS ≤ 1) were included. The patients were grouped and analyzed according to reversed shock index < 1 or reversed shock index ≥ 1.
  Interventions: Other: reversed shock index < 1; Other: reversed shock index ≥ 1

INTERVENTIONS:
Other: reversed shock index < 1 — Among patients with isolated TBI, those with an RSI < 1 had higher mortality
Other: reversed shock index ≥ 1 — Among patients with isolated TBI, those with an RSI ≥ 1 had lower mortality

SUMMARY:
A systolic blood pressure (SBP) lower than the heart rate (HR) could indicate a poor condition in trauma patients. In such scenarios, the reversed shock index (RSI) is <1, as calculated by the SBP divided by the HR. This study aimed to clarify whether RSI could be used to identify high-risk adult patients with isolated traumatic brain injury (TBI).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients having isolated TBI with a head abbreviated injury scale (AIS) ≥ 3 and without severe injury to other regions (other AIS ≤ 1) were included

Exclusion Criteria:

* Patients with incomplete registered data were also excluded

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients having isolated TBI with a head abbreviated injury scale (AIS) ≥ 3 and without severe injury to other regions (other AIS ≤ 1) were included. We excluded patients younger than 18 or older than 65 years of age. Patients were grouped and analyzed according to RSI (< 1 or ≥ 1).
Sampling Method: Probability Sample
Enrollment: 1216 (Actual)
Dates: Start 2016-03-23 (Actual); Primary Completion 2017-01-23 (Actual); Study Completion 2017-02-22 (Actual)

PRIMARY OUTCOMES:
in-hospital mortality | up to 5 months
  To measure the outcome of patients.

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data available.